CLINICAL TRIAL: NCT02791672
Title: Perioperative Care of Breast Reconstruction With Latissimus Dorsi Flap and Tissue Expander: Early Discharge Protocol in a Day Surgery Setting
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Jing Zhang, Staff Plastic Surgeon, University of Ottawa
Other Study IDs: 20160216-01H
Record Dates: First submitted 2016-05-31; First posted 2016-06-07 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-05

CONDITIONS: Mammaplasty
Keywords: Perioperative Care; Breast Reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Same Day Discharge: Following a Latissimus Dorsi flap reconstruction patients will be offered discharge at 24 hours. Patients successfully discharged within 24 hours of their surgery will be included in the cohort group.
  Interventions: Behavioral: Discharge within 24 hours

INTERVENTIONS:
Behavioral: Discharge within 24 hours — If both the physician and patient have no concerns within 24 hours of a Latissimus Dorsi Flap breast reconstruction the patient will be discharged home and enrolled in the cohort group.

SUMMARY:
The pedicled latissimus dorsi flap is a piece of tissue taken from the back that is used to reconstruct the breast after cancerous tissue is removed. Over the years, improvements in surgical technique and pain control have decreased the length of stay in hospital after this procedure. Recently, early discharge after breast reconstruction using another very similar pedicled flap, called the transverse rectus abdominis flap, was shown to be safe, patient-centered, and associated with significant hospital cost-savings by another Canadian group.

With increasing pressure from hospital administrators to weigh financial considerations into treatment decision making, doctors must test cost-saving strategies in order to ensure patient satisfaction and safety. Here, we plan to evaluate patient safety, satisfaction and cost efficacy in breast reconstruction using the pedicled latissimus dorsi myocutaneous flap.

We hypothesize that patient care planning can allow for safe and cost-effective same-day discharge and improved patient satisfaction after autologous breast reconstruction using the pedicled latissimus dorsi flap. After nearly 10 successful same-day discharges using this flap, our experience at the Ottawa Hospital suggests that this practice is safe, has increased patient satisfaction scores, decreased narcotic use, no short or long term complications and is more cost effective compared to patients who stay overnight.

In the present study, we hope to quantify our results by demonstrating that same day discharge is a cost effective strategy that does not compromise patient safety and satisfaction.

DETAILED DESCRIPTION:
The pedicled latissimus dorsi myocutaneous flap is a reliable option for autologous breast reconstruction after mastectomy. Improvements in technique and postoperative analgesia have decreased the length of hospital stay required after this procedure. Early discharge following a range of procedures has been consistently shown to increase patient satisfaction, decrease perioperative complication rates, and improve hospital cost-effectiveness. Specifically, early discharge after breast reconstruction using another pedicled myocutaneous flap, the transverse rectus abdominis myocutaneous flap, was shown to be safe, patient-centered, and associated with significant hospital cost-savings by another Canadian group.

The balance between financial savings and patient safety/comfort has been studied vigorously across many medical disciplines. With increasing pressure from hospital administrators to weigh financial considerations into treatment decision making, clinicians must empirically test cost-saving strategies in order to ensure patient satisfaction and safety.

Here, we evaluate patient safety, satisfaction and cost efficacy in ambulatory breast reconstruction using the pedicled latissimus dorsi myocutaneous flap.

ELIGIBILITY:
Inclusion Criteria:

* All patients who undergo breast reconstruction using the latissimus dorsi myocutaneous flap.

Exclusion Criteria:

* All patients undergoing breast reconstruction without the latissimus dorsi flap.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be females older than 18 years old who undergo breast reconstructive surgery with the Latissimus Dorsi flap.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Conversion rate (from same-day discharge to in-patient care) | 24 hours
Patient Satisfaction using Breast-Q questionnaire and Perioperative Care Patient | 24 hours
Pain Score | 24 hours
Amount of post-operative (24 hours) narcotic usage | 24 hours

SECONDARY OUTCOMES:
Short and Long term complications | 24 Hours
Readmission Rate | 24 Hours
Cost Savings | 24 Hours

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will not be made available. Anonymity will be maintained for all published data.